CLINICAL TRIAL: NCT06236009
Title: A Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled, Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of TAK-004 in Healthy Subjects
Brief Title: A First-In-Human Study of TAK-004 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: TAK-004-1001
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: TAK-004 or Placebo (Single Ascending Dose Cohorts) (Experimental): Participants will receive TAK-004 or matching-placebo subcutaneous injection on Day 1 in Cohort S1 using a sentinel dosing scheme in a double-blind manner. After dosing the first two participants in Cohort S1, the investigator will review all available safety and tolerability data up to 24 hours post-dose before dosing the remaining participants in the Cohort S2-S10. Single ascending doses are nominal and may be modified based on emerging safety and available PK data during the study but will have a corresponding dose that does not exceed the maximal defined exposure.
  Interventions: Drug: TAK-004; Drug: Placebo
- Part 2: TAK-004 or Placebo (Multiple Ascending Dose Cohorts) (Experimental): Participants will receive TAK-004 (dose to be decided [TBD]) or matching-placebo subcutaneous injection, once daily for 5 days (i.e., Day 1 to 5) in each 5 multi-ascending dose cohorts (M1-M5). The dose in Part 2 will be determined at the dose escalation meeting based upon emerging safety, tolerability, and available PK data from Part 1.
  Interventions: Drug: TAK-004; Drug: Placebo
- Part 3: TAK-004 or Placebo (Expansion Cohorts) (Experimental): Participants will receive TAK-004 (TBD) or matching-placebo subcutaneous injection on Day 1 in each single ascending dose expansion cohorts (E1 and E2). Doses will be determined at the dose escalation meeting based on safety, tolerability and available PK data from Parts 1 and 2. Expansion cohort 2 (optional) may be conducted at the sponsor's discretion after reviewing expansion cohort 1 data.
  Interventions: Drug: TAK-004; Drug: Placebo

INTERVENTIONS:
Drug: TAK-004 — TAK-004 subcutaneous injections.
Drug: Placebo — Matching- placebo subcutaneous injections.

SUMMARY:
This study is the first study with TAK-004 conducted in human beings. Participants will receive either TAK-004 or placebo. The main aim of this study is to learn how safe TAK-004 is in healthy adults and how well participants tolerate one or more doses of TAK-004. Other aims are to learn about the effects of TAK-004 on the heart rate and blood pressure and if TAK-004 creates an immune response (immunogenicity). Another aim is to learn how the body of healthy adults affects TAK-004 (pharmacokinetics).

Participants will receive TAK-004 or placebo via injection just under the skin (subcutaneous injection or SC injection). Depending on the groups participants are assigned to, they will either receive just one dose of TAK-004 or placebo or multiple doses of TAK-004 or placebo while they are in the study. Blood and urine samples will be taken during the study.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for participation in this study, the participant must:

1. Understand the study procedures and agree to participate by providing written informed consent.
2. Be willing and able to comply with all study procedures and restrictions and follow all rules and regulations while confined in the clinical research unit.
3. Be a healthy male or woman of nonchildbearing potential (WONCBP) participant aged 18 to 55 years, inclusive, at the screening visit.
4. Continuous nonsmoker who has not used nicotine- and tobacco-containing products for at least 3 months before dosing.
5. Has not had frequent or heavy use (i.e., near-daily) of medical or recreational cannabis for at least 3 months before screening.
6. Has a body mass index greater than or equal to (>=) 18 and less than or equal to (<=) 30.0 kilogram per square meter (kg/m^2) at the screening visit.
7. Be judged to be in good health (example, no evidence of psychiatric, hepatic, renal, pulmonary, or cardiovascular disease) by the investigator, based on clinical evaluations including laboratory safety tests, medical history, physical examination, ECG, and vital sign measurements performed at the screening visit and before administration of the initial dose of IP or invasive procedure.
8. Meet the following birth control requirements:

   * Is a male participant who is sterile or agrees to use an appropriate method of contraception, including a condom with or without spermicidal cream or jelly, from the first dose of IP until 5 half-lives after the last dose of IP. No restrictions are required for a vasectomized male participant provided the participant is at least 4 months after bilateral vasectomy procedure before the first dose of IP. A male participant whose vasectomy procedure was performed less than 4 months before the first dose of IP must follow the same restrictions as a non-vasectomized man. Appropriate documentation of surgical procedure should be provided.
   * Is a male participant who agrees not to donate sperm from the first dose of IP until 5 half-lives after the last dose of IP.
   * Is a WONCBP, defined by at least 1 of the following criteria:

     1. Postmenopausal (defined as 12 months of spontaneous amenorrhea in females aged greater than (>) 45 years or 6 months of spontaneous amenorrhea in females aged >45 years with serum follicle-stimulating hormone (FSH) levels >40 milli-international units per milliliter [mIU/mL]). Appropriate documentation of FSH levels is required.
     2. Surgically sterile by hysterectomy and/or bilateral oophorectomy with appropriate documentation of surgical procedure.
     3. Had a bilateral tubal ligation, bilateral tubal occlusion, or bilateral salpingectomy with appropriate documentation of surgical procedure.
     4. Has a congenital condition resulting in no uterus.

Exclusion Criteria:

Any participant who meets any of the following criteria will not qualify for entry into the study:

1. The participant has participated in another investigational study within 4 weeks (or based on local regulations) or within 5 half-lives of the IP before the day of check-in. The 4-week or 5 half-lives window will be derived from the date of the last IP administration and/or AE related to the IP administration in the previous study to the day of check-in of the current study.
2. The participant is an employee of the sponsor or study site or immediate family member (example, spouse, parent, child, sibling) of the sponsor or study site.
3. The participant has a history of significant multiple and/or severe allergies (example, food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerance to prescription or nonprescription drugs or food. A history of mild seasonal allergies/allergic rhinitis is allowed at the investigator's discretion.
4. The participant has a known hypersensitivity or contraindication to any component of TAK-004.
5. The participant has a positive pregnancy test result or is lactating or breastfeeding.
6. The participant has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency antibody/antigen, at the screening visit.
7. The participant had major surgery or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks before the screening visit.
8. The participant is unable to refrain from or anticipates using medications including herbal medicines beginning approximately 7 days before administration of the first dose of IP.
9. The participant is unable to refrain from or anticipates using marijuana or cannabis-containing products from screening, through check-in (Day -2) or within 15 days of drug administration (whichever is longer).
10. The participant has a history or presence of alcoholism or drug abuse within the past 2 years before dosing.
11. The participant drinks alcohol in excess of 21 glasses/units per week for males or 14 glasses/units per week for females, with one unit = 150 mL of wine or 360 mL of beer or 45 mL of 45% alcohol.
12. Positive alcohol test result at check in, or positive urine drug screen results at screening or check-in.
13. The participant has a history of major psychotic disorder.
14. The participant has a history or presence of:

    * Cardiovascular Exclusion:

      * 2 or more incidences of vasovagal syncope within the last 5 years before screening;
      * A family history of unexplained sudden death or channelopathy;
      * Brugada syndrome (ie, RBBB pattern with ST-elevation in leads V1-V3);
      * Cardiovascular or cerebrovascular disease, such as cardiac valvulopathy, myocardial infarction, stroke, sick sinus syndrome, pulmonary congestion, any cardiac arrhythmias (including ventricular tachycardia), second-degree AV block type 2, third-degree AV block, prolonged QT interval with Fridericia correction method (QTcF) interval, hypokalemia, hypomagnesemia, or conduction abnormalities;
      * Risk factors for Torsade de Pointes (eg, heart failure, cardiomyopathy, or family history of Long QT Syndrome);
      * Any clinically significant ECG findings or medical history including long or short QT interval with Fridericia correction method (QTcF) (over 450 millisecond [msec] or less than 360 msec), bifascicular block, left anterior hemiblock/fascicular block or QRS >=120 msec or PR interval >210 msec from screening to Day 1 pre-dose (inclusive);
      * A documented history or at screening/check-in of sinus bradycardia (<55 beats per minute [bpm]), sinoatrial block or sinus pause >=3 seconds.
    * Renal Disease Exclusion:

      * Any relevant personal or family history of renal disease.
      * Any clinically significant elevation of blood urea nitrogen or serum creatinine and/or an abnormal glomerular filtration rate.
      * Urinalysis finding suggestive of kidney injury.
15. The participant has an average semi-recumbent BP less than 90/60 millimeter of mercury (mmHg) or greater than 140/90 mmHg from screening to Day 1 pre-dose, inclusive. Any assessments on Day -1, where 2 consecutive time point values do not meet this criterion, will be exclusionary.
16. The participant has an average HR <55 or >100 bpm from screening to Day 1 pre-dose, inclusive. Any assessments after admission with an average HR <55 bpm or HR >100 bpm, from Day -2 to Day 1 pre-dose (inclusive), will be left to the judgment of the investigator, where 2 consecutive time point values do not meet this criterion, the participant will not be eligible.
17. The participant has orthostatic hypotension defined as a decrease in SBP >=20 mm Hg or a decrease in DBP >=10 mm Hg at approximately 3 minutes of standing when compared with BP from the semi-recumbent position at screening to Day 1 pre-dose assessments, inclusive. In asymptomatic participants, any assessments that do not meet this criterion may be repeated after the participant has remained in the semi-recumbent or supine position for at least 15 minutes. If the repeat assessment is exclusionary based on the above criterion, the participant will not be eligible. If the repeat assessment is not exclusionary, the participant will be eligible.
18. The participant has postural orthostatic tachycardia, defined as an increase of >30 bpm or HR >120 bpm at approximately 3 minutes of standing, at screening to Day 1 pre-dose assessments, inclusive. Any assessments that do not meet this criterion may be repeated with the participant remaining standing for up to a total of 5 minutes, provided that the participant remains asymptomatic. If the repeat assessment occurring within 5 minutes is exclusionary based on the above criterion, the participant will not be eligible.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | From the first dose of study drug up to 60 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study investigational product (IP), whether or not the occurrence is considered related to the study IP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of the study IP. An untoward finding generally may necessitate therapeutic intervention, require an invasive diagnostic procedure, or require discontinuation or a change in dose of IP or a concomitant medication. Any clinically significant vital signs, electrocardiogram (ECG)/telemetry/Holter monitoring, laboratory values will be considered as AEs.

SECONDARY OUTCOMES:
Orthostatic Changes in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Values From Semi-Recumbent to Standing at 0.5 Hours After First Dose | From semi-recumbent to standing at 0.5 hours after first dose (Day 1)
Changes in Semi-Recumbent Heart Rate (HR) Values at 2 Hours After First Dose | At 2 hours after first dose (Day 1)
Number of Participants with Antidrug Antibody (ADA) Status | From the first dose of study drug up to 60 days
  The number participants in each category of the ADA status (ADA-negative or ADA-positive) will be determined in this study. A 3-tiered ADA testing strategy will be used in this study. A Sample will initially be screened for ADA by the ADA screening assay. Any positive sample in the screening assay is considered a potential positive, which will be confirmed for true positivity by the confirmatory assay. If a sample is confirmed as an ADA true positive, ADA titer will be assessed.
Parts 1 and 2: Maximum Observed Plasma Concentration (Cmax ) for TAK-004 | Part 1: Pre-dose (Day 1), 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, 24, 30, 48, 72 and 96 hours post-dose; Part 2: Pre-dose (Day 1), 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, and 24 hours at Days 1 and 5 post-dose
Part 1: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-inf) for TAK-004 | Part 1: Pre-dose (Day 1), 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, 24, 30, 48, 72 and 96 hours post-dose
Parts 1 and 2: Time to Reach the Maximum Plasma Concentration (Tmax) for TAK-004 | Part 1: Pre-dose (Day 1), 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, 24, 30, 48, 72 and 96 hours post-dose; Part 2: Pre-dose (Day 1), 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, and 24 hours at Days 1 and 5 post-dose
Part 1: Area Under the Plasma Concentration-Time Curve From Time 0 To Time of The Last Quantifiable Concentration (AUC0-last) for TAK-004 | Part 1: Pre-dose (Day 1), 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, 24, 30, 48, 72 and 96 hours post-dose
Parts 1 and 2: Terminal Disposition Phase Half-life (T1/2z) for TAK-004 | Part 1: Pre-dose (Day 1). 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, 24, 30, 48, 72 and 96 hours post-dose; Part 2: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, and 24 hours post-dose at Day 5
Parts 1 and 2: Apparent Clearance After Extravascular Administration (CL/F) for TAK-004 | Part 1: Pre-dose (Day 1). 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, 24, 30, 48, 72 and 96 hours post-dose; Part 2: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, and 24 hours post-dose at Day 5
Parts 1 and 2: Apparent Volume of Distribution During the Terminal Disposition Phase After Extravascular Administration (Vz/F) for TAK-004 | Part 1: Pre-dose (Day 1). 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, 24, 30, 48, 72 and 96 hours post-dose; Part 2: Pre-dose, 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, and 24 hours post-dose at Day 5
Part 2: Area Under the Plasma Concentration-time Curve From Time 0 to tau Over Dosing Interval (AUCtau) for TAK-004 | Part 2: Pre-dose (Day 1), 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, and 24 hours post-dose at Days 1 and 5
Part 2: Observed Plasma Concentration at the end of a Dosing Interval (Ctrough) for TAK-004 | Part 2: 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, and 24 hours post-dose at Day 5
Part 2: Accumulation Ratio Based on AUCtau (Rac[AUC]) After a Single Dose for TAK-004 | Part 2: 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, and 24 hours post-dose at Day 5
  Rac(AUC) will be calculated as AUCtau on Day 5 divided by AUCtau after a single dose.
Part 2: Accumulation Ratio Based on Cmax (Rac[Cmax]) for TAK-004 | Part 2: 0.25, 0.5, 1, 2, 3, 4, 5, 7, 10, 14, and 24 hours post-dose at Day 5
  Rac(Cmax) will be calculated as Cmax on Day 5 divided by Cmax after a single dose.
Parts 1 and 2: Amount of Drug Excreted in Urine From Time 0 to Time t (Aet) for TAK-004 | Part 1: Pre-dose, 0-7, 7-12 and 12-24 hours post-dose at Day 1; Part 2: Pre-dose, 0-7, 7-12 and 12-24 hours post-dose at Days 1 and 5
Parts 1, 2: Amount of Drug Excreted in Urine From Time 1 to Time 2 (Aet1-t2) for TAK-004 | Part 1: Pre-dose, 0-7, 7-12 and 12-24 hours post-dose at Day 1; Part 2: Pre-dose, 0-7, 7-12 and 12-24 hours post-dose at Days 1 and 5
Parts 1 and 2: Amount of Drug Excreted in Urine During a Dosing Interval (Aeτ) at Steady State for TAK-004 | Part 1: Pre-dose, 0-7, 7-12 and 12-24 hours post-dose at Day 1; Part 2: Pre-dose, 0-7, 7-12 and 12-24 hours post-dose at Days 1 and 5
Parts 1 and 2: Fraction of Administered Dose of Drug Excreted From Urine From Time 0 to Time t (fe,t) for TAK-004 | Part 1: Pre-dose, 0-7, 7-12 and 12-24 hours post-dose at Day 1; Part 2: Pre-dose, 0-7, 7-12 and 12-24 hours post-dose at Days 1 and 5
Parts 1 and 2: Renal Clearance (CLR) for TAK-004 | Part 1: Pre-dose, 0-7, 7-12 and 12-24 hours post-dose at Day 1; Part 2: Pre-dose, 0-7, 7-12 and 12-24 hours post-dose at Days 1 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/256f8c1e888a4fef??page=1&idFilter=TAK-004-1001